CLINICAL TRIAL: NCT07053358
Title: An Exploratory Clinical Study Evaluating LX111 Gene Therapy in Patients With Neovascular Age-related Macular Degeneration (nAMD)
Brief Title: Safety and Efficacy Evaluation of LX111 Gene Therapy in nAMD Patients
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: Innostellar Biotherapeutics Co.,Ltd (Industry)
Responsible Party: Principal Investigator, Xiaodong Sun, PhD, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHGH-LX111
Record Dates: First submitted 2025-06-27; First posted 2025-07-08 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Neovascular Age-related Macular Degeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LX111 intravitreal injections (Experimental)
  Interventions: Genetic: LX111 Injection

INTERVENTIONS:
Genetic: LX111 Injection — Qualified subjects will receive a single unilateral intravitreal injection of LX111 at Day 0.

SUMMARY:
The goal of this study is to evaluate the safety and efficacy of LX111 treatment of nAMD. This study will enroll subjects aged ≥ 50 vears old to receive a single unilateral intravitreal (lVT) injection of LX111 to evaluate its safety and efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Willing to sign the informed consent, and willing to attend follow-up visits.
2. Age ≥ 50
3. Diagnosis of active CNV secondary to neovascular AMD
4. BCVA ETDRS letters between 5 and 63
5. Subjects must have received a minimum of 2 injections within 6 months prior to screening and demonstrated a meaningful response to anti-VEGF therapy
6. Male subjects whose partner is a fertile female or female subjects who are fertile, agree to take effective contraceptive measures from the screening period until the last follow-up.

Exclusion Criteria:

1. CNV or macular edema in the study eye secondary to diseases other than nAMD
2. Retinal detachment, uveitis, uncontrolled glaucoma in the study eye, or any condition preventing visual acuity improvement
3. Acute coronary syndrome, myocardial infarction or coronary artery revascularization, CVA, TIA in the last 6 months
4. Uncontrolled hypertension defined as average SBP ≥160 mmHg or an average DBP ≥100 mmHg
5. Uncontrolled diabetes defined as HbA1c >8.0% within 28 days prior to screening

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-07-02 (Estimated); Primary Completion 2026-11-23 (Estimated); Study Completion 2029-12-30 (Estimated)

PRIMARY OUTCOMES:
Adverse events and serious adverse events in the eyes and throughout the body within 364 days after LX111 treatment | 52 weeks
  Incidence of adverse events and serious adverse events within 52 weeks of LX111 intravitreal injection in each dose group.
Dose Limiting Toxicity | 4 weeks
  The incidence of DLT in each dose group.

SECONDARY OUTCOMES:
Mean changes in BCVA from Baseline | 12 weeks, 36 weeks, 52 weeks
  The mean changes of BCVA scores on the ETDRS chart at different timepoints after LX111 treatment compared with baseline.
Mean changes in Central Subfield Thickness (CST) from Baseline | 12 weeks, 36 weeks, 52 weeks
  The mean changes of CST at different timepoints after LX111 treatment compared with baseline.
The percentage of subjects who received anti-VEGF supplemental injection within 52 weeks after LX111 treatment | 52 weeks
  The proportion of subjects who received anti-VEGF supplemental injection within 52 weeks after LX111 treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, China

IPD SHARING:
Plan to Share IPD: No